CLINICAL TRIAL: NCT06667427
Title: Pilot Study of Management of Facial Paralysis in the Oncologic Patient: Nerve Transfer Techniques to Improve Facial Function and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1315; NCI-2024-09091 (Other: NCI-CTRP Clinical Trials Registray)
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Head and Neck Cancer
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Participants will be identified and recruited during their visit to the Center of Reconstructive Surgery.
  Interventions: Procedure: Nerve transfer techniques
- Surgery (Experimental)
  Interventions: Procedure: Nerve transfer techniques

INTERVENTIONS:
Procedure: Nerve transfer techniques — Participants will undergo facial nerve reconstruction using nerve transfer techniques

SUMMARY:
The goal of this research study is to measure changes in patients' quality of life after surgeries that affect the facial nerve, including nerve transfer as treatment for facial paralysis.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the impact of facial nerve transfer techniques (FNTT) on QoL in head and neck cancer patients with facial paralysis. This study intends to measure the impact of FNTT on QoL utilizing a series of validated questionnaires which include: (i) Facial Clinimetric Evaluation Scale and Facial Disability Index; (ii) Sunnybrook Facial Grading System; and (iii) Facial Nerve Grading Scale 2.0. These instruments will be administered at baseline, after surgery, and at 6, 12, and 18 months post-operatively.

Secondary Objective:

To compare patient-reported outcomes and facial function scales for patients who undergo facial nerve transfer technique with a historical cohort of patients who did not undergo any dynamic nerve reconstruction procedures. The same assessment tools described in primary objective above will be utilized.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in the intervention group of this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form
* Aged 18 or greater
* Patient scheduled to undergo facial nerve transfer
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study

In order to be eligible to participate in the non-intervention historical control group of this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form
* Aged 18 or greater
* Previous facial surgery severing a facial nerve without graft or other form of dynamic facial nerve reconstruction within the last 5 years

Exclusion Criteria:

Patients known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Z-Hye Lee, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org